CLINICAL TRIAL: NCT00001285
Title: Chronobiologic Effects of Gonadal Steroid Manipulations in Volunteer Subjects
Brief Title: Effects of Sex Hormones on Circadian Rhythm in Men and Women
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 910206; 91-M-0206
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-10

CONDITIONS: Bipolar Disorder; Circadian Rhythm; Depressive Disorder
Keywords: Circadian Rhythms; Environmental Light; Estrogen; Melatonin; Progesterone; Rapid Cycling Bipolar Disorder; Sleep; Testosterone; Depression; Hypomania; Mania
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder; Depression; Mania

SUMMARY:
For many years researchers have been trying to better understand the regulation of sleep and activity by studying circadian (daily) rhythms of human beings. It appears that the hormones estrogen, progesterone, and testosterone play a role in the regulation of circadian rhythm in animals. Researchers believe these hormones may also play a similar role in the regulation of human circadian rhythms. Little research has been conducted on how these hormones affect human circadian rhythms.

This study is designed to learn more about how specific hormones influence men and women's daily rhythms. This study will use women from another research study being conducted at the NIMH called, "The central nervous system effects of pharmacologically induced hypogonadotropic hypogonadism with and without estrogen and progesterone". Male subjects will be recruited from another NIMH study called, "The central nervous system effects of pharmacologically induced hypogonadotropic hypogonadism with and without testosterone replacement".

In order to test the possibility that gonadal steroids (estrogen, progesterone, and testosterone) change circadian rhythms and the sleep-wake cycle in humans, participants will undergo chronobiologic evaluations. The chronobiologic evaluations will look at sleep and rest periods, activity as measured by a wrist monitor, and 24 hour inpatient electroencephalograph (EEG), rectal temperature, and melatonin monitoring.

DETAILED DESCRIPTION:
It is hypothesized that gonadal steroids modulate circadian rhythms and the sleep-wake cycle in humans, as they do in animals. This hypothesis will be tested by performing chronobiologic evaluations on women enrolled in protocol 92-M-0174 ("The central nervous system effects of pharmacologically induced hypogonadotropic hypogonadism with and without estrogen and progesterone") and on men enrolled in protocol 94-M-0037 (The central nervous system effects of pharmacologically induced hypogonadotropic hypogonadism with and without testosterone replacement"). Based on the animal literature, we hypothesize that melatonin and sleep onset will be phase-advanced in women on estrogen, compared with those on progesterone or in a hypogonadal state. We also hypothesize that the amplitude of the activity cycle will be decreased in the progesterone, as compared with the estrogen, condition. Based on findings in amenorrheic women and in those on oral contraceptives, we hypothesize that the amplitude of melatonin secretion will be increased in the hypogonadal state, compared with the other two conditions. Finally, based on literature cited below, we hypothesize that mean prolactin levels will be higher in the testosterone plus Lupron condition and in the estrogen plus Lupron condition than in the other hormonal conditions.

ELIGIBILITY:
Volunteers must be healthy individuals between the ages of 18 and 45 years old.

No pregnant women.

No history of menstrually-related mood or behavioral disturbances.

No volunteers with current or past Axis I diagnoses, significant abnormalities on physical or neurological examination, or significant laboratory abnormalities.

Must be HIV negative.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 73
Dates: Start 1991-08; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Leibenluft E. Do gonadal steroids regulate circadian rhythms in humans? J Affect Disord. 1993 Oct-Nov;29(2-3):175-81. doi: 10.1016/0165-0327(93)90031-e. PMID 8300976
- [Background] Leibenluft E, Schmidt PJ, Turner EH, Danaceau MA, Ashman SB, Wehr TA, Rubinow DR. Effects of leuprolide-induced hypogonadism and testosterone replacement on sleep, melatonin, and prolactin secretion in men. J Clin Endocrinol Metab. 1997 Oct;82(10):3203-7. doi: 10.1210/jcem.82.10.4270. PMID 9329339
- [Background] Albers HE. Gonadal hormones organize and modulate the circadian system of the rat. Am J Physiol. 1981 Jul;241(1):R62-6. doi: 10.1152/ajpregu.1981.241.1.R62. PMID 7246802